CLINICAL TRIAL: NCT06884501
Title: Let's Increase Fuerza (Strength) Through Exercise and Diet
Acronym: LIFTED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Susan Aguinaga, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB24-1409
Record Dates: First submitted 2024-11-19; First posted 2025-03-19 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Older Adults (50-90 Years); Cognition; Physical Activity
Keywords: strength training; Latinos; Latin dance; physical activity; cognition; brain health; dietary pattern
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Remote-delivered BAILAMOS™ dance program, MIND diet & strength training
  Interventions: Behavioral: Latin dance, MIND diet, and Strength training
- Control Group (Active Comparator): Remote-delivered BAILAMOS™ dance program and MIND diet
  Interventions: Behavioral: Latin dance and MIND Diet

INTERVENTIONS:
Behavioral: Latin dance, MIND diet, and Strength training — This will be a 6 month remote-delivered BAILAMOS™ dance program, MIND diet and strength training intervention.
  Arms: Intervention Group
Behavioral: Latin dance and MIND Diet — This will be a 6 month remote-delivered BAILAMOS™ dance and MIND diet program.
  Arms: Control Group

SUMMARY:
The purpose of the study is to conduct a 6-month randomized controlled trial among Latinos ages 50+ at risk for cognitive decline and compare the efficacy of a remote-delivered, culturally tailored Latin dance program and strength training coupled with a Mediterranean-Dash Intervention for Neurodegenerative Delay (MIND) diet (IG) compared to a Latin dance and MIND diet program (CG) on cognitive performance, CVD risk factors, MIND diet adherence, physical activity, biomarkers, and psychosocial outcomes.

Participants will:

* Randomly be placed in the intervention (IG) or control group (CG)
* Have 2 pre and post intervention testing visits
* Have weekly sessions during the 6-month trial

DETAILED DESCRIPTION:
Screening and Consent: Potential participants can consent to be screened via email or by calling our office to be screened. Study staff will screen all interested individuals for eligibility based on inclusion/exclusion criteria. Participants will be administered the Exercise and Screening for You (EASY) tool. The EASY tool consists of 6 questions to assess one's risk factors associated with exercise. Depending on how participants respond to the 6 questions, they may need to obtain medical clearance to participate in the study.

To obtain medical clearance, we will ask interested participants for the name and contact information of physician. We will send a letter via email or fax to the physician requesting medical clearance. Once we receive medical clearance vi email or fax, we will then begin the Informed Consent process. Once determined eligible, study staff will email Qualtrics link to Informed Consent and will go over the consent form. Participants will be instructed to save/print a copy of the document for their records. After participants have signed the Informed Consent, they will be invited to the first testing session at Freer Hall at the University of Illinois at Urbana-Champaign.

Baseline first testing session (~2 hours): At the first testing session, research personnel will collect demographics, health history, self-reported physical activity (Godin & non-exercise measure of cardiorespiratory fitness), and the Food Frequency Questionnaire will be administered. Anthropometrics such as height, weight, blood pressure, waist circumference, and DEXA scan will also be conducted.

Trained research staff will guide the participant through drop sets (increasing weight with decreasing repetitions) with 10 reps (2lbs), 8 reps (3lbs), 6 reps (5lbs), and 4 reps (8lbs) for the following exercises: Dumbbell overhead press, dumbbell squat, dumbbell single arm row, dumbbell deadlift, seated dumbbell chest fly, and dumbell side lunges. We will have participants begin with light weights and slowly progress with heavier weights (if possible, otherwise participants will stick to lighter weights). These exercise have been chosen for the baseline and posttesting because they are reflective of the exercise that they wil do at home.

Participants will be provided with an accelerometer and the accelerometer log. Participants will be asked to wear the accelerometer for 7 consecutive days. Participants will be asked to wear the monitor on a belt or attached to a clip placed on their non-dominant hip during wake times only. They will be asked to remove the monitor during any water-related activities and sleep. Accelerometer-wearing instructions and logs will be provided to participants. After the 7 days, participants will be scheduled for their second visit.

Randomization: Participants will be randomly assigned to one of two groups after participants complete the first baseline visit: 1) intervention group (IG) remote-delivered BAILAMOS™ dance program, MIND diet & strength training; or 2) control group (CG) remote-delivered BAILAMOS™ dance program and MIND diet. Participants in the IG group will meet 3 times a week for a total of 4 hrs per week and the CG will meet twice week for 3 hrs per week.

Baseline second testing session (~2 hours): At the second testing session, vegetable consumption will be assessed through the Veggie Meter. In brief, the Veggie Meter is a non-invasive device that measures vegetable consumption through LED lighting. Participants are asked to insert their non-dominant ring finger into the scanner and a carotenoid score between 0-800 is provided to participant. A cognitive battery will also be administered. A set of psychosocial questionnaires (NIH Toolbox Perceived Stress, General Life Satisfaction, Sadness, and Loneliness) will also be administered. Given that this is a remote-delivered intervention, participants will then be instructed to download Zoom to their computer or iPad device (they will be asked to bring these devices). Research staff will provide participants with an e-mail with a LIFTED study ID. Additionally, research staff will help participants troubleshoot through Zoom, if needed. Participants in the IG will be provided with resistance bands and two sets of weights (5lb and 10lb weights) for the strength training program.

Interventions:

Remote-delivered BAILAMOS™ dance program: BAILAMOS™ is a Latin dance, Spanish-language intervention that encompasses six dance styles. The program meets twice weekly for 60 minutes per session during 6-months. It encompasses six dance styles: Merengue, Cha Cha Cha, Bachata, Salsa, Cumbia and Flamenco. The instructor will follow a specific protocol containing a step-by-step guide of each dance class. It will be delivered via Zoom. A trained dance instructor (with 5+ years of dance instruction experience) with experience in leading dance classes for older adults will deliver the dance sessions. Each session will begin with reviewing safety procedures, stepping in place as a warm-up, followed by stretching. Instruction begins with the basics of the respective styles of dance, followed by advanced steps for singles. Over each month, activity increases and progresses in terms of movement, specificity of dance moves, and complexity. Basic principles are targeted, such as partnership, timing, footwork, and movement quality. Each session ends with a 5-minute cool-down. Logs will assess the rate of perceived exertion and heart rate. Participants will completes these via paper logs. They will receive 6-months worth of log sheets during baseline testing visit 2. Participants will be reminded to increase their lifestyle PA.

Remote-delivered MIND Diet program: The Mediterranean-DASH diet intervention for neurodegenerative delay (MIND) is a diet that is tailored for the protection of the brain and contains the most compelling evidence of reduction of dementia. The MIND diet consists of 10 brain-healthy food groups (green leafy vegetables, other vegetables, nuts, berries, beans, whole grains, seafood, poultry, olive oil, and wine). The MIND diet also recommends a limited intake of foods that are unhealthy for the brain (high saturated fat or sugar intakes, such as red meat and meat products, butter, whole-fat cheese, pastries and sweets, and fried/fast foods). The intervention group will receive one MIND diet session per week. The MIND Diet program will be delivered via Zoom in a group discussion setting by a trained graduate student with a background in nutrition (Bachelor's degree in nutrition or current training in nutrition). The instructor will follow a specific study protocol that contains information on all sessions. The first 30 minutes of the session will introduce the food item, describe its benefits, and describe ways to incorporate these food items into their diet. During this portion, the instructor will make participants aware of any allergy concerns related to the food items that are introduced. The second half of the session (30 minutes) will consist of culturally appropriate recipes, food demonstrations, and recipe sharing by both instructors and participants.

Remote delivered strength training program: The IG will receive a two 30 minute strength group training sessions led by an ACSM certified personal trainer. The program includes a twice a week session of 30-minutes, delivered over 6-months and is group-based. The study-specific strength training protocol consists of three sets of 8-12 repetitions of six different resistance exercises targeting all major muscle groups. Participants will begin with bodyweight and progress to use 5lbs, and if possible, 10lbs weights. Instructions will be provided on proper form. Exercises include Dumbbell overhead press, dumbbell squat, dumbbell single arm row, dumbbell deadlift, seated dumbbell chest fly, and dumbell side lunges however, exercises may be modified to accommodate participant's physical abilities. Each session will end with a 5-minute cool-down.

All sessions will be recorded, and stored in a secure server. Participants will be invited to make-up missed sessions using the recorded videos. These will be completed on a one-on-one basis with a trained researcher.

Post-testing: All participants will then be asked to participate in the 6-month post-intervention testing sessions (2 testing sessions). All tests will be administered in the same order at baseline and month 6 testing. Each participant will have three weeks to complete testing, thus we may test participants at month 6+3 weeks. After that, participants will not be allowed to be tested for the 6-month testing.

Post-testing first testing session (~2 hours): The pre and post surveys will be linked via participant ID numbers. At the first testing session, research personnel will collect anthropometrics such as height, weight, blood pressure, waist circumference, and DEXA scan. Self-reported physical activity questionnaires will be administered (Godin & non-exercise measure of cardiorespiratory fitness). Trained research staff will guide the participant through drop sets (increasing weight with decreasing repetitions) with 10 reps (2lbs), 8 reps (3lbs), 6 reps (5lbs), and 4 reps (8lbs) for the following exercises: Dumbbell overhead press, dumbbell squat, dumbbell single arm row, dumbbell deadlift, seated dumbbell chest fly, and dumbell side lunges.

Participants will be provided with an accelerometer and the accelerometer log. Participants will be asked to wear the accelerometer for 7 consecutive days. Participants will be asked to wear the monitor on a belt or attached to a clip placed on their non-dominant hip during wake times only. They will be asked to remove the monitor during any water-related activities and sleep. Accelerometer-wearing instructions and logs will be provided to participants. After the 7 days, participants will be scheduled for their second visit.

Post-testing second testing session (~2 hours): At second testing session, the Food Frequency Questionnaire will be administered. A set of psychosocial questionnaires (NIH Toolbox Perceived Stress, General Life Satisfaction, Sadness, and Loneliness) will also be administered. Vegetable consumption will be assessed through the Veggie Meter. The Veggie Meter measures vegetable and fruit consumption using light spectroscopy. Participants are asked to insert their non-dominant ring finger into the scanner and a carotenoid score between 0-800 is provided to participants. A cognitive battery will also be administered.

ELIGIBILITY:
Inclusion Criteria:

1) self-identify as a Latino/Hispanic, 2) age 50+, 3) documented cardiovascular disease (CVD) or at least one CVD risk factor (i.e., hypertension, hyperlipidemia, diabetes, obesity, current smoker, or family history of CVD), 3) participate in <3 days or <90 minutes of moderate-to-vigorous PA per week, 4) able to understand Spanish, 5) Wi-Fi Access, 6) score of greater than 21 on the TICS-M

Exclusion Criteria:

1. uncontrolled illness including diabetes (e.g., participant reports high glucose levels despite treatment efforts), hypertension (e.g., participant is hypertensive while on medication or not adhering to medication), or thyroid disease (e.g., patient reports experiencing hyperthyroidism).
2. history of musculoskeletal, cardiorespiratory, or neurological diseases that preclude the participation in moderate intensity exercise

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Stroop Neuropsychological Screening Test (Trennerry et al., 1989) | Change in score from baseline to 6 months
  Stroop Test will be used to assess executive function. In Stroop C, participants are shown a list of colors printed in conflicting color ink and are asked to read words (names of colors). The second part of this task is Stroop CW in which participants are shown a list of colors printed in conflicting color ink and are asked to say the color of the ink the word is printed. The scores are the number of words named correctly in 30 seconds and the number of colors named correctly in 30 seconds subtracting the number of errors. respectively.
Word fluency Test (Welsh et al., 1994) | Change in score from baseline to 6 months
  Word Fluency will be used to assess executive function. The Word Fluency Test asks participants to name as many animals (part 1) or fruits and vegetables (part 2) as possible in 60 seconds. The score is the sum of the number of animals and the number of fruits and vegetables named.
Digit Span Test (Wechsler, 1987) | Change in score from baseline to 6 months
  Digit Span Test will be used to measure executive function. Digit Span Forward & Backward will be used to assess working memory. Digit strings of increasing length will be read, and the participant is asked to repeat each string forward (Digit Span Forward) or backward (Digit Span Backward). The score is the number of correctly retrieved strings in each part
Trail Making Test (A&B) | Change in scores from baseline to post-intervention 6 months
  Trail Making Test (A&B) will be used to measure executive function. Part A consists of numbers spread out in a grid with a dedicated start and end point. Participants must trace in sequential order. Part B will consist of numbers and letters in sequential order spread across a grid with a start and end point as well. Participants much trace the starting number to letter. Scoring will be based on seconds needed to complete each test with Part A having a max of 100 seconds and Part B with a max of 300 seconds. Test will discontinue when the time limit has been reached.

SECONDARY OUTCOMES:
Minutes per day of light and moderate-to-vigorous physical activity via GT3x Actigraph Accelerometer | Change in minutes per day of light and moderate-to-vigorous physical activity from baseline to post-intervention 6 months
  Device-assessed physical activity via GT3x Actigraph accelerometers will be used to assess minutes per day spent in light physical activity and moderate-to-vigorous physical activity.
Godin-Shephard Leisure-Time Physical Activity Questionnaire | Change in score from baseline to 6 months
  The Godin-Shephard Leisure-Time Physical Activity Questionniare is 2-item questionnared used to assess leisure time physical activity.
Non-exercise Cardiorespiratory Fitness Questionnare | Change in score from baseline to 6 months
  The non-exercise cardiorespiratory fitness questionnaire estimates cardiorespiratory fitness using age, sex, BMI, resting heart rate, and self-reported physical activity.
Spectroscopy-Based Veggie Meter® | Change in scores from baseline to post-intervention 6 months
  The Veggie Meter (VM; Longevity Link Inc., Salt Lake City, UT, USA) is a commercially available device that uses reflection spectroscopy to measure the level of carotenoid pigments in a person's skin by scanning the tip of the finger. Scores range from 0-800.
Plasma Structural Lipidomics | Change in scores from baseline to post-intervention 6 months
  A lipidomics profile will be assessed from the plasma provided. This will be analyzed with Liquid Chromatography coupled to Mass Spectrometry to identify over 800 lipid species
National Institutes of Health (NIH) Toolbox: Perceived Stress Fixed Form Age 18+ v2.0 | Change in scores from baseline to post-intervention 6 months
  NIH Tool box measure of perceived stress is a self-reported measure that assesses how unpredictable, uncontrollable, and overloaded respondents find their lives. 10 items are administered using a 5-point scale, with options ranging from "never" to "very often". Higher scores are indicative of higher perceived stress.
National Institutes of Health (NIH) Toolbox General Life Satisfaction Fixed Form A Age 18+ v2.0 | Change in scores from baseline to post-intervention 6 months
  NIH Tool box measure of general life satisfaction assesses global feelings and attitudes about one's life. 5 items are administered using a 5 and 7-point scale, ranging from "strongly disagree" to "strongly agree". Higher scores are indicative of higher general life satisfaction.
National Institutes of Health (NIH) Tool Box: Sadness Fixed Form Age 18+ v2.0 | Change in scores from baseline to post-intervention 6 months
  NIH Toolbox measure of depression/sadness assesses negative mood, negative views of self, and negative social cognition. 8 items are administered using a 5-point scale ranging from "never" to "always". Higher scores are indicative of more sadness.
National Institues of Health (NIH) Toolbox Loneliness Fixed Form Age 18+ v2.0 | Change in scores from baseline to post-intervention 6 months
  NIH Toolbox measure of loneliness assesses perceptions of loneliness using 5 items, responses from a 5-point scale ranging from "never" to "always". Higher scores are indicative of more loneliness.
MIND Diet Adherence | Change in scores from baseline to post-intervention 6 months
  Block 2005 Food Frequency Questionnaire will be used to compute MIND diet scores. Frequency of consumption for food items was assigned a score of 0, 0.5, or 1, where scores ranged from 0 (lowest adherence) to 15 (highest adherence)
Blood pressure | Change from baseline to post-intervention 6 months
  Blood pressure will be assessed using Omron blood pressure monitors
Fasting Blood glucose | Change from baseline to post-intervention 6 months
  2, 3 mL blood samples will be obtained to assess fasting blood glucose.
Waist Circumference | Change from baseline to post-intervention 6 months
  Waist circumference will be measured using a tape measure reported as CM.
DEXA | Change from baseline to post-intervention 6 months
  A DEXA scan is a type of x-ray that will be used used to measure body composition.
MOCA-Blind Version 8.1 | Change in score from baseline to 6 months
  The MOCA-Blind assesses attention, concentration, memory, language, conceptual thinking, calculations, and orientation.

IPD SHARING:
Plan to Share IPD: Undecided